CLINICAL TRIAL: NCT06339138
Title: Identification of Novel High Quality Methylated DNA Markers in Renal Tumors: Whole Methylome Discovery, Tissue Validation, and Feasibility Testing in Blood and Urine
Brief Title: Identification of Novel High Quality Methylated DNA Markers in Renal Tumors: Whole Methylome Discovery, Tissue Validation, and Feasibility Testing In Blood and Urine, The INQUIRE Study
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-010944; NCI-2024-00971 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-010944 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chromophobe Renal Cell Carcinoma; Clear Cell Papillary Renal Tumor; Clear Cell Renal Cell Carcinoma; Kidney Oncocytoma; Papillary Renal Cell Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Oncocytoma, renal; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples retained with permission of participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants may undergo blood, urine, and tissue sample collection on study. Participants' medical records are also reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to collect blood, tissue and urine samples to identify a novel high quality methylated DNA marker in patients with renal tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In tissue, to discover and validate DNA methylation markers (MDMs) for detection of malignant renal and urothelial tumors.

II. In blood, to assess the accuracy of candidate MDMs from above for detection of malignant renal and urothelial tumors.

OUTLINE: This is an observational study.

Participants may undergo blood, urine, and tissue sample collection on study. Participants' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* CASE TISSUE:

  * Patient has a histological diagnosis of primary clear cell RCC, papillary cell RCC, clear cell papillary RCC, chromophobe RCC, oncocytoma, or urothelial cell carcinoma
  * Age >= 18 years
* CASE BLOODS AND URINE:

  * Patient has a histological diagnosis of primary clear cell RCC, papillary cell RCC, chromophobe RCC, oncocytoma, or urothelial cell carcinoma
  * Age >= 18 years
* HEALTHY CONTROL BLOODS AND URINE:

  * Patients has undergone negative hematuria workups (defined as negative abdominal imaging and negative cystoscopy
  * Age >= 18 years

Exclusion Criteria:

* CASE TISSUE:

  * Patient has von Hippel-Lindau disease (VHL), Hereditary leiomyomatosis and renal cell cancer (HLRCC), Hereditary papillary renal carcinoma (HPRC), or Birt-Hogg-Dube syndrome (BHD)
  * The current target pathology is a recurrence
  * Patient has undergone any prior radiation therapy to target lesion prior to surgery
  * Patient has received chemotherapy class drugs in the 5 years prior to surgery
  * Patient has had any transplants prior to surgery
  * Patient has confirmation of Lynch Syndrome, is presumed to have Lynch Syndrome, or has familial cancer syndrome X
  * Patient has Nephritis (Glomerulus or Interstitial), Poly Cystic Kidney Disease, Glomerulonephropathies or Acquired Renal Kidney Disease
* RENAL CONTROL TISSUE:

  * Patient has von Hippel-Lindau disease (VHL), Hereditary leiomyomatosis and renal cell cancer (HLRCC), Hereditary papillary renal carcinoma (HPRC), or Birt-Hogg-Dube syndrome (BHD).
  * Patient has inflammation, atypia, or hyperplasia of the parenchyma
  * Patient has a current or past history of renal cancer.
  * Patient has undergone any prior radiation therapy to target lesion prior to surgery
  * Patient has received chemotherapy class drugs in the 5 years prior to surgery
  * Patient has had any transplants prior to surgery
  * Patient has confirmation of Lynch Syndrome, is presumed to have Lynch Syndrome, or has familial cancer syndrome X
  * Patient has Nephritis (Glomerulus or Interstitial), Poly Cystic Kidney Disease, Glomerulonephropathies or Acquired Renal Kidney Disease
* UROTHELIAL CONTROL TISSUE:

  * Patient has von Hippel-Lindau disease (VHL), Hereditary leiomyomatosis and renal cell cancer (HLRCC), Hereditary papillary renal carcinoma (HPRC), or Birt-Hogg-Dubé syndrome (BHD)
  * Patient has inflammation, atypia, or hyperplasia of the urothelium
  * Patient has a current or past history of urothelial cancer
  * Patient has undergone any prior radiation therapy to target lesion prior to surgery
  * Patient has received chemotherapy class drugs in the 5 years prior to surgery
  * Patient has had any transplants prior to surgery
  * Patient has confirmed or presumed lynch
* CASE BLOODS AND URINE:

  * Patient has known primary cancer outside of the kidney within the last 5 years prior to plasma and urine collection (not including basal cell or squamous cell skin cancers)
  * Patient has had surgery to completely or partially remove current target pathology
  * Patient has undergone any prior radiation therapy to target lesion prior to plasma and urine collection
  * Patient has received chemotherapy class drugs in the 5 years prior to plasma and urine collection
  * Patient has had any transplants prior to plasma and urine collection
  * Patient has confirmed or presumed lynch
  * Patient has von Hippel-Lindau disease (VHL), Hereditary leiomyomatosis and renal cell cancer (HLRCC), Hereditary papillary renal carcinoma (HPRC), or Birt-Hogg-Dubé syndrome (BHD)
* HEALTHY CONTROL BLOODS AND URINE:

  * Patient has known primary cancer outside of the urothelium within the last 5 years prior to plasma and urine collection (not including basal cell or squamous cell skin cancers)
  * Current target pathology is a recurrence
  * Patient has undergone prior radiation therapy in the 5 years prior to plasma and urine collection
  * Patient has received chemotherapy class drugs in the 5 years prior to plasma and urine collection
  * Patient has had any transplants prior to plasma and urine collection
  * Patient has von Hippel-Lindau disease (VHL), Hereditary leiomyomatosis and renal cell cancer (HLRCC), Hereditary papillary renal carcinoma (HPRC), or Birt-Hogg-Dube syndrome (BHD)
  * Patient has confirmed or presumed lynch
  * Gross urinary incontinence
  * Patient has undergone cystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a histological diagnosis of primary clear cell RCC, papillary cell RCC, clear cell papillary RCC, chromophobe RCC, oncocytoma, urothelial cell carcinoma, or healthy participants who have undergone negative hematuria workups
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Identify novel methylated DNA markers in tissue for malignant renal and urothelial tumors | Baseline (at enrollment)
  Assessed by the number of markers identified using unbiased whole methylome sequencing (RRBS). Top candidates will be validated in independent tissue. Potential markers will have relatively low background and a false discovery rate 20%.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Kisiel, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials